CLINICAL TRIAL: NCT00193141
Title: Paclitaxel, Carboplatin, Infusional 5-Fluorouracil, and Radiation Therapy With or Without Surgical Resection in Locally Advanced Esophageal Cancer
Brief Title: Chemotherapy With or Without Surgical Resection in Locally Advanced Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: SCRI Oncology Research Consortium, SCRI
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 23
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Esophagus Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel; Carboplatin; Fluorouracil

INTERVENTIONS:
Drug: Paclitaxel
Drug: Carboplatin
Drug: 5-Fluorouracil

SUMMARY:
In this randomized study, we plan to address the important question of optimum local treatment for patients with localized esophageal cancer. All patients will receive our previously studied neo-adjuvant regimen including paclitaxel, carboplatin, infusional 5-FU, and radiation therapy to 45 Gy. At the completion of neo-adjuvant therapy, patients will be randomized to undergo surgical resection, or to continue radiation to a total dose of 60 Gy, along with one additional course of chemotherapy.

DETAILED DESCRIPTION:
Upon determination of eligibility, all patients will receive neo-adjuvant therapy with:

Paclitaxel + Carboplatin + 5-Fluorouracil + Radiation

After neo-adjuvant therapy and restaging are completed, patients will be randomized to receive one of two treatments:

* Surgical resection (Arm A)
* Paclitaxel + Carboplatin + Radiation (Arm B)

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Cancer of the esophagus or gastroesophageal junction confirmed by biopsy (squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma) clinical stage I, II, or III.
* Received no previous treatment for esophageal cancer.
* Measurable or evaluable disease
* Able to perform activities of daily living with minimal assistance
* Adequate bone marrow, liver and kidney function
* Be at least 3 weeks from any major surgical procedures.
* Have an indwelling central venous access catheter.
* Patients must be able to understand the nature consent of the study and give written informed consent.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Age < 18 years
* History of a prior malignancy within the past 5 years
* History of significant heart disease
* Inoperable on the basis of co-existent medical problems

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 1999-10; Primary Completion 2004-10 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of full dose radiation therapy versus preoperative radiation therapy plus surgical resection, when used in combination with neo-adjuvant chemotherapy, in the treatment of localized esophageal cancer

SECONDARY OUTCOMES:
To compare the toxicity of these two treatment approaches in localized esophageal cancer
To evaluate the utility of clinical restaging in guiding local therapy (surgical resection vs definitive radiation therapy) following neo-adjuvant treatment
To evaluate the toxicity of additional chemotherapy and radiation therapy following completion of neo-adjuvant treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Result] Hainsworth JD, Meluch AA, Gray JR, Spigel DR, Meng C, Bearden JD, Hermann R, Greco FA. Concurrent chemoradiation followed by esophageal resection vs chemoradiation alone for localized esophageal cancer. Community Oncology 4:431-439, 2007.
- See also: Community Oncology article — http://www.communityoncology.net/journal/articles/0407431.pdf